CLINICAL TRIAL: NCT04631874
Title: A Phase 1 Clinical Trial to Compare and Evaluate Safety and Pharmacokinetic Characteristics After Administration of the "CDFF0318" and "Champix Tab. 1mg (Varenicline Tartrate)" in Healthy Male Volunteers
Brief Title: A Clinical Trial to Compare Pharmacokinetics of the "CDFF0318" and "Champix Tab. 1mg"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTC Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTC-IND-CDFF0318_1
Record Dates: First submitted 2020-10-27; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Smoking Cessation; Pharmacokinetics
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A(RT) (Experimental): Reference drug (Champix) -> washout -> test drug (CDFF0318)
  Interventions: Drug: CDFF0318, Champix
- Sequence B(TR) (Experimental): Test drug (CDFF0318) -> washout -> reference drug (Champix)
  Interventions: Drug: CDFF0318, Champix

INTERVENTIONS:
Drug: CDFF0318, Champix — CDFF0318: Varenicline salt changed Champix: Varenicline tartrate

SUMMARY:
A Phase 1 Clinical Trial to Compare and Evaluate Safety and Pharmacokinetic Characteristics after Administration of the "CDFF0318" and "Champix Tab. 1mg (Varenicline tartrate)" in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 19 to 45 years
* a body mass index of 18.0-30.0 kg/m2

Exclusion Criteria:

* Subjects with disease history or current disease of clinically significant liver, kidney, nervous system, respiratory system, endocrine system, blood/tumor, urinary system, cardiovascular system, etc.
* Subjects with a history of gastrointestinal diseases or gastrointestinal surgery that may affect the absorption of investigational drugs
* Subjects with a history of hypersensitivity reactions or clinically significant hypersensitivity reactions to drugs containing varenicline and other drugs (ketoprofen, aspirin, antibiotics, etc.)
* Subjects who have an abnormal diet that may affect the absorption, distribution, metabolism, and excretion of the drug, or who eat food that may affect drug metabolism

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (AUC0-t) | 72 hours
  AUC0-t of "CDFF0318" and "Champix Tab. 1mg"
Pharmacokinetics (Cmax) | 72 hours
  Cmax of "CDFF0318" and "Champix Tab. 1mg"

SECONDARY OUTCOMES:
Safety and tolerability (Vital sign) | 72 hours
  Blood pressure (mmHg)
Safety and tolerability (Vital sign) | 72 hours
  Heart rate (beats/min)
Safety and tolerability (12-lead ECG) | 72 hours
  ventricular rate (beats/min)
Safety and tolerability (12-lead ECG) | 72 hours
  PR interval (msec)
Safety and tolerability (Laboratory tests) | 72 hours
  Creatinine [mg/dL]
Safety and tolerability (Laboratory tests) | 72 hours
  AST, ALT [IU/L]
Safety and tolerability (Laboratory tests) | 72 hours
  eGFR [mL/min/1.73m^2]
Safety and tolerability (Adverse events) | 72 hours
  Adverse events were collected regardless of the time point when the subject complained of symptoms.
  Adverse events were assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Min-Kyu Park, Principal Investigator — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No